CLINICAL TRIAL: NCT07207226
Title: Arterial Stiffness as a Tool to Investigate Adherence in Resistant Hypertension
Acronym: INSIDE-RH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C23-84; IDRCB (Registry Identifier: 2024-A00270-47)
Record Dates: First submitted 2025-01-08; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Resistant Hypertension (Experimental): Participants with resistant hypertension defined as - - Blood pressure at consultation > 140 and/or 90 mmHg and/or 24h-ABPM (Ambulatory Blood Pressure Assessment) and/or in Home blood pressure measurement (HBPM) > 130 and/or 80 mmHg despite taking three or more different classes of antihypertensive drugs at optimal doses, including a diuretic, on the day of screening irrespective of the BP on the day of the visit.
  - Any office BP, ABPM or HBPM values in patients taking four or more different classes of antihypertensive drugs at optimal doses, including a diuretic.
  Interventions: Device: Laser doppler vibrometry

INTERVENTIONS:
Device: Laser doppler vibrometry — Non-invasive CARDIS Technology Demonstrator (CTD) device is a 2 x 6 beam laser Doppler vibrometer (LDV) for non-contact measurement of skin vibrations caused by underlying cardiac action. The CTD device is a split device with a master device and a slave device, which are connected to a data acquisition rack, which again is connected to a computer for signal processing, data presentation and data logging.

SUMMARY:
According to WHO estimates, worldwide, 1.28 billion adults between the age of 30-79 years have hypertension. Furthermore, only 1 in 5 people with hypertension have it under control. In approximately 15% of the patients treated for hypertension, optimum blood pressure levels are not achieved even after the addition of 3-4 conventional anti-hypertensive drugs. These patients are diagnosed as resistant hypertensives. Resistant hypertension is associated with an increased risk of cardiovascular death, myocardial infarction, and stroke.

Hypertension is a chronic condition where arterial pressures are persistently elevated, leading to an increase in the pulsatile load on the arteries. This can result in structural and functional alterations in the arterial wall leading to an increase in 'arterial stiffness'.

Arterial stiffness is dependent on the mechanical load (blood pressure) and the material properties of the vessel wall. There is a vicious loop between hypertension and arterial stiffness, where hypertension may lead to alteration in the vascular structure and cause degradation of the elastic components of the vessel wall, and an increase in arterial stiffness can lead to higher blood pressure. An increase in arterial stiffness is associated with higher cardiovascular disease (CVD) risk, and patients with resistant hypertension are at a significantly higher risk of developing CVD. Measurement of carotid-femoral pulse wave velocity (PWV) is considered the gold standard for assessing arterial stiffness and has been recommended as a method to evaluate arterial stiffness as a part of routine care in patients with hypertension. The European Society of Hypertension (ESH) and the working group of the European Society of Cardiology (ESC) recommend its use for the evaluation of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-90 years of age in both sexes, diagnosed with resistant hypertension.
* - Resistance Hypertension defined as -
* Blood pressure at consultation > 140 and/or 90 mmHg and/or 24h-ABPM (Ambulatory Blood Pressure Assessment) and/or in Home blood pressure measurement (HBPM) > 130 and/or 80 mmHg despite taking three or more different classes of antihypertensive drugs at optimal doses, including a diuretic, on the day of screening irrespective of the BP on the day of the visit.
* Any office BP, ABPM or HBPM values in patients taking four or more different classes of antihypertensive drugs at optimal doses, including a diuretic.
* Patients scheduled for arterial stiffness assessment as a part of routine treatment.
* Patients eligible or affiliated with a social security scheme.
* Patients who provide written informed consent for participation.

Exclusion Criteria:

* - Inability to express consent to the study
* Persons subject to a judicial safeguard measure, under guardianship or curatorship.
* Patients with skin lesions (severe eczema, wounds, etc.) on the chest or neck that do not allow the application of the protective skin film on the area of interest; Allergies to the adhesive film.
* Subjects not affiliated with social security or an equivalent scheme.
* Linguistic incapacity or psychic refusal to read the information.
* Diseases carrying out a life -expectancy <1 year according to clinical judgment
* Pregnant women (because of physiological hemodynamic changes in BP and stiffness during pregnancy)
* Arrhythmias: current AC/FA, high degree BAV.
* Persons subject to a period of exclusion for another research
* Foreseen inability to attend scheduled visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Measurement of Carotid-femoral PWV (Pulse wave velocity) by applanation tonometry using a Sphygmocor device | Baseline and Between 20 and 24 weeks after the baseline visit
  The technique is non-invasive and will be made with the patient in a supine position. This measurement is repeated three times to ensure accuracy according to international recommendations

SECONDARY OUTCOMES:
Measurement of heart-carotide PWV (Pulse Wave Velocity) by LDV (Laser Doppler Vibrometer) | Baseline and Between 20 and 24 weeks after the baseline visit
  The measurement will be taken from the neck (carotid) to the groin (femoral) site
Measurement of antihypertensive drug concentration | Baseline and Between 20 and 24 weeks after the baseline visit
  Drug levels will be tested in routine urine samples.
Categorize adherence phenotype | Baseline and Between 8 and 16 weeks after the baseline visit
  Urine samples will be taken on a dried matrix

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Georges pompidou, Paris, Île-de-France Region, France